CLINICAL TRIAL: NCT02464436
Title: First-in-human Phase I/IIa, Open-Label, Prospective Study of the Safety and Tolerability of Subretinally Transplanted Human Retinal Progenitor Cells (hRPC) in Patients With Retinitis Pigmentosa (RP)
Brief Title: Safety and Tolerability of hRPC in Retinitis Pigmentosa
Acronym: hRPCRP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ReNeuron Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN03-CP-0001
Record Dates: First submitted 2015-05-18; First posted 2015-06-08 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Retinitis Pigmentosa
Keywords: RP
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- human retinal progenitor cells (hRPC) (Experimental): Single subretinal administration of human retinal progenitor cells (hRPC)
  Interventions: Drug: hRPC

INTERVENTIONS:
Drug: hRPC — Participants will undergo vitrectomy surgery and subretinal implantation of hRPC in the study eye.
  Other Names: human retinal progenitor cells

SUMMARY:
hRPC is a cell therapy for retinitis pigmentosa. This is a first-in-human, dose escalation study in which participants with retinitis pigmentosa will receive a single subretinal injection of hRPC cells in one eye to evaluate safety and tolerability.

Participants will be followed for two years to evaluate the safety and tolerability of hRPC Additional testing will seek to establish any preliminary efficacy from hRPC.

DETAILED DESCRIPTION:
This is a first-in-human open label phase I/II dose-escalation study in which participants with retinitis pigmentosa will receive a single uni-ocular subretinal implantation of one of three doses of hRPC.

Treated eyes will be carefully monitored for any ocular or systemic adverse events for 2 years.

Testing will comprise a series of detailed ophthalmic examinations and imaging together with blood testing and systemic evaluations, as necessary.

Ophthalmic testing will also be evaluated for any preliminary efficacy signal.

ELIGIBILITY:
Inclusion Criteria:

1. Have ability to give written informed consent as evidenced by signature on the subject consent form.
2. Be adult male or female over 18 years of age.
3. Have clinical diagnosis of RP, based upon one or more of the following: clinical features, medical imaging, electrophysiological measures and genetic testing, if available. Genetic confirmation is not obligatory.
4. Have Best Corrected ETDRS visual acuity of 35 letters or less (approximately 20/200 or worse) in the study eye for cohorts 1-5; have Best Corrected ETDRS visual acuity of 63 letters (approximately 20/63) to 36letters (approximately 20/200) in the study eye for cohorts 6-8, and Best Corrected ETDRS visual acuity of 8 letters (approximately 20/800) to 68 letters (approximately 20/50) for cohorts 9 and on.
5. Be able to complete the entire microperimetry test, and demonstrate adequate fixation and consistency between baseline readings such that the accuracy of both baseline and follow on testing should enable the detection of clinically significant changes in retinal sensitivity.
6. Be medically able to undergo vitrectomy and subretinal injection.
7. Have good general health as defined by:

   * Normal serum chemistry and hematology. Out of normal range laboratory findings deemed not clinically significant are acceptable.
   * No history of malignancy, except non-melanoma skin cancer; pre-malignant conditions and cancer in situ.
   * Negative serology for human immunodeficiency virus (HIV), hepatitis B (HBV), hepatitis C (HCV).
   * Medically fit enough to undertake surgery which may require general anesthesia as well as medically fit to undergo a short perioperative course of systemic corticosteroid therapy
   * Free of any other systemic condition that in the opinion of the Investigator may have an impact on the safety of the subject, conduct of study procedures, or integrity of study data (e.g. severe cardiovascular or respiratory disease; poorly controlled diabetes; significant psychiatric impairment).
8. Females of childbearing potential must have a confirmed negative pregnancy test at Visits 1 and 3; and be willing to use highly effective method of contraception (e.g. oral contraceptive and condom, intra-uterine device (IUD) and condom, diaphragm with spermicide and condom) for the duration of this study.
9. Males must be willing to use a reliable method of contraception (e.g. barrier and spermicide) for the duration of this study; unless have been surgically sterilized with confirmed azoospermia.
10. Be willing and able to attend all scheduled clinical assessments, ability to communicate well with the Investigator and to comply with the expectations of the study.

Exclusion Criteria:

1. Exhibits a difference in ETDRS BCVA of 15 letters of more in either eye between any of the baseline visits.
2. Exhibits a difference in ETDRS BCVA of 20 or more letters between eyes at the time of any of the screening or baseline visits attributed to asymmetry in the progression of RP.
3. Presence of ocular disease or ocular media opacity in the study eye, which in the opinion of the Investigator, will preclude an accurate evaluation at any time during the study.
4. History of any retinal and/or macular disease other than RP (e.g. retinal detachment) that in the opinion of the Investigator may have an impact on the safety of the subject, conduct of study procedures, or integrity of study data.Specifically, subjects in whom significant pre-existing vitreoretinal pathology might influence visual acuity outcomes should be excluded
5. Active ocular infection or inflammation, or any history of intraocular inflammation, that would expose subject to risk during or following surgery.
6. Prior vitrectomy in the study eye.
7. A history of amblyopia in the study eye.
8. High myopia (>6 diopters) in the study eye.
9. Cataract surgery in the study eye or ocular surgery in either eye (which in the opinion of the investigator may have an impact on patient safety or the integrity of data from the study eye) during the study or within 3 months prior to treatment.
10. Participation in any clinical study involving an investigational drug or device within 6 months prior to treatment or 5 half-lives of the drug (whichever is longer) prior to initiation of treatment
11. Prior stem cell administration or injections to any part of the body (subjects who have received autologous bone marrow stem cell transplant will be eligible).
12. Use of systemic immunosuppressive agents (e.g. corticosteroid) in the 6 months prior to treatment or 5 half-lives of the drug (whichever is longer) prior to initiation of treatment (Note: inhaled, intranasal, and/or topical dermatologic steroids are allowed)
13. (For females) Be breastfeeding or planning a pregnancy.

m) Known hypersensitivity to any of ingredients of the excipient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12; Primary Completion 2022-06 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety over the six months after treatment as assessed by the incidence of treatment emergent adverse events (TEAEs) and changes from baseline in other safety parameters. | 6 months
  Safety measures will be assessed by review of important events, including but not limited to inflammation, complications of the surgical procedure and worsening of vision.

SECONDARY OUTCOMES:
Safety (Visual function measure: change in visual acuity) | 24 months
  A summary of the ETDRS +/- BRVT BCVA letter score and the change from baseline to end of study in the treated eye presented by treatment group.
Safety (Visual function measure: change in visual field: Goldmann visual field, microperimetry and FST) | 24 months
  A summary of the perimetry and change from baseline to end of study in the treated eye presented by treatment group.
Safety (Change in retinal sensitivity in the area overlying the implanted hRPC as compared with untreated retina) | 24 months
  ERG results and change from baseline to end of study summarized descriptively and presented by treatment group.
Safety (Anatomical endpoint relating to retinal function in implant location - Color Fundus Photography) | 24 months
  A qualitative description of the change in retinal appearance of treated and untreated retinal area in the treated eye from baseline to end of study presented by treatment group.
Safety (Anatomical endpoint relating to retinal function in implant location - Fundus autofluorescence) | 24 months
  A qualitative description of the change in retinal appearance of treated and untreated retinal area in the treated eye from baseline to end of study presented by treatment group.
Safety (Anatomical endpoint relating to retinal function in implant location - Spectral domain-OCT) | 24 months
  Summary of the overall retinal thickness, outer nuclear layer thickness and ellipsoid zone measurement and change from baseline to the end of study of treated retina compared with untreated retina in the treated eye by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Comander, MD, Principal Investigator — Massachusetts Eye and Ear Infirmary (MEEI); Vince Holmes, Study Director — ReNeuron Limited
Locations (5):
- United States (3):
  - Retinal Research Institute, Phoenix, Arizona
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Oregon Health and Science University, Portland, Oregon
- Institut de la Màcula, Barcelona, Spain
- Oxford Eye Hospital, Oxford, United Kingdom